CLINICAL TRIAL: NCT05535504
Title: Multi-center, Prospective, Comparative, Randomized, Double Blind, Superior, Pivotal Study to Compare and Evaluate the Efficacy and Safety of Repetitive Transcranial Magnetic Stimulation Applied With an Electromagnetic Therapy Stimulator 'ALTMS-A' for Upper-limb Motor Function Recovery With the Sham Control Group for Those Who Need Upper-limb Rehabilitation Treatment for Subcortical and Brainstem Stroke (Ischemic)
Brief Title: The Efficacy & Safety of rTMS for Upper-limb Motor Function Recovery in Subcortical and Brainstem Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty in patient recruitment
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-2205-756-001
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Hemiplegia; Subcortical Infarction
Keywords: Stroke; Transcranial magnetic stimulation; Rehabilitation; Neuronal plasticity; Subcortical infarction
MeSH Terms: conditions — Stroke; Hemiplegia; Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: ALTMS-A
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real rTMS (Experimental): Use the real rTMS coil
  Interventions: Device: Low-frequency rTMS (experimental)
- sham rTMS (Sham Comparator): Use the sham rTMS coil
  Interventions: Device: Low-frequency rTMS (sham comparator)

INTERVENTIONS:
Device: Low-frequency rTMS (experimental) — Frequency: Low-frequency (1Hz) rTMS / Intensity: 100% of resting motor threshold / Location: motor hotspot of the contralesional primary motor cortex (the first dorsal interosseous muscle) / Number of total stimuli : 1800 ; Coil orientation: tangential to scalp
  Arms: real rTMS
Device: Low-frequency rTMS (sham comparator) — Frequency: Low-frequency (1Hz) rTMS / Intensity: 100% of resting motor threshold / motor hotspot of the contralesional primary motor cortex (the first dorsal interosseous muscle) / Number of total stimuli : 1800 ; Coil orientation: vertical to scalp
  Arms: sham rTMS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of repetitive transcranial magnetic stimulation applied with an electromagnetic therapy stimulator 'ALTMS-A' for upper-limb motor function recovery with the sham control group for those who need upper-limb rehabilitation treatment for subcortical and brainstem stroke

DETAILED DESCRIPTION:
After low-frequency repetitive transcranial magnetic stimulation (rTMS) over the contralesional motor cortex (M1), the score of the Box and Block test increased immediately, especially in patients without cortical involvement.

Eighty-eight patients will be recruited and divided into two groups. Each group will receive 10 sessions of the real rTMS or sham rTMS over the contralesional primary motor cortex. Each rTMS session consists of low-frequency (1Hz) 1800 stimulations.

The objective of this study is to evaluate the efficacy and safety of rTMS for upper-limb motor function in patients with subcortical and brainstem stroke.

ELIGIBILITY:
Inclusion Criteria:

* 19-80 years old
* Radiologically confirmed ischemic stroke with subcortical and brainstem lesions within 90 days
* Fugl-Meyer assessment scale (upper extremity) > 15
* Mini-mental status exam (the Korean version) > 14 with appropriate cognitive function
* Written informed consent

Exclusion Criteria:

* Fugl-Meyer assessment scale (wrist) < 1 or Fugl-Meyer assessment scale (hand) < 1
* Hemorrhagic stroke or traumatic brain injury
* Cerebellar stroke
* Previous history of stroke
* Traumatic brain injury
* Previous history of brain surgery
* Need for intensive care due to complications associated with stroke (e.g. pneumonia, infection, hemodynamic instability)
* History of psychological or neurological diseases
* History of pain or muscular weakness of upper limbs which may interfere with rehabilitation
* History of seizure or epilepsy
* Aphasia
* Skin lesions in the stimulation site of scalp
* Intracranial metal implant
* Inability to receive regular physical or occupational therapy
* Disagreement to use contraception in women of childbearing age

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Box and Block test | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS

SECONDARY OUTCOMES:
Box and Block test | upto 14 days
  Before rTMS (baseline) and immediately after the completion of 10 sessions of rTMS
Fugl-Meyer Assessment Scale | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
modified Barthel Index (the Korean version) | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
National Institutes of Health Stroke Scale | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
Finger tapping | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
Brunnstrom stage (hand and arm) | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
Modified Ashworth scale (wrist flexor, wrist extensor, elbow flexor, elbow extensor, and finger flexor) | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS
Grip strength (hand grip, pinch grip, lateral prehension, three jaw chuck) | upto 42 days
  Before rTMS (baseline) and 4 weeks after the completion of 10 sessions of rTMS

OTHER OUTCOMES:
Vital sign | upto 42 days
  Before rTMS (baseline), immediately after the completion of 10 sessions of rTMS, and 4 weeks after the completion of 10 sessions of rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (2):
- South Korea (2):
  - Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do
  - Department of Rehabilitation Medicine, Chungnam National University Hospital, Korea, Daejeon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho HM, Cha S, Sohn MK, Jee S, Chang WK, Kim WS, Paik NJ. Investigation of the efficacy of low-frequency repetitive transcranial magnetic stimulation on upper-limb motor recovery in subacute ischemic stroke without cortical involvement: a protocol paper for a multi-center, double-blind randomized controlled trial. Front Neurol. 2023 Aug 25;14:1216510. doi: 10.3389/fneur.2023.1216510. eCollection 2023. PMID 37693768